CLINICAL TRIAL: NCT01451970
Title: Assessing the Effects of Two Diets Enriched in Either Saturated or Unsaturated Fatty Acids to Determine the Cellular and Molecular Mechanisms in Insulin Sensitivity
Brief Title: Dietary Fatty Acid Composition and Obesity-related Metabolic Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Robert C. Atkins Foundation (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N009310
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Overweight/Obese Women
Keywords: high fat diet treatment; insulin sensitivity
MeSH Terms: conditions — Overweight; Insulin Resistance | interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Monounsaturated Fat Diet (Other): Subjects will adhere to their specific diet for four weeks. The diet will be a weight-maintaining diet, and the target nutrient composition for diets will be 55% carbohydrate, 30% fat, 15% protein. For the monounsaturated fat treatment (M diet) approximately 10% of all lipids ingested will be saturated.
  Interventions: Other: High Fat Diet
- High Saturated Fat Diet (Other): Subjects will adhere to their specific diet for four weeks. The diet will be a weight-maintaining diet, and the target nutrient composition for diets will be 55% carbohydrate, 30% fat, 15% protein. For the saturated fat treatment (S diet) approximately 40% of all lipids ingested will be saturated.
  Interventions: Other: High Fat Diet

INTERVENTIONS:
Other: High Fat Diet — Subjects will adhere to their specific diet for four weeks. For both diet treatments, the diet will be a weight-maintaining diet, and the target nutrient composition for diets will be 55% carbohydrate, 30% fat, 15% protein. For the monounsaturated fat treatment (M diet) approximately 10% of all lipids ingested will be saturated. For the saturated fat treatment (S diet) approximately 40% of all lipids ingested will be saturated.

SUMMARY:
Individuals have a significant capacity to adapt to different environments by changing their core metabolic pathways. This adaptation is especially important in regards to diet. Epidemiological research over the last several decades have shown that diets high in saturated fats have a greater ability to cause insulin resistance and the 'metabolic syndrome' while diets low in saturated fats (or a so called 'Mediterranean Diet), reduces the risk for cardiovascular disease. In humans, experimental diets high in unsaturated fats, as compared to high carbohydrate or high saturated fat diets, result in increased insulin sensitivity and improved lipid profiles.

In this application, the investigators propose to systematically assess the effects of two diets enriched in either saturated or unsaturated fatty acids and determine the cellular and molecular mechanisms of the apparent increase in insulin sensitivity. The investigators hypothesize that individuals will 'adapt' to the different diets and the investigators will be able to generate predictive alterations in gene expression and metabolites that underlie the alterations in metabolism. In parallel, the investigators will test the ability of these different diets to affect the release of gastrointestinal hormones that may be critical to modulation of appetite.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females with BMI range of 25-32 kg/m2

Exclusion Criteria:

* Evidence of metabolic or cardiovascular disease, Fasting plasma glucose concentration > 125mg/dl, Abnormal EKG, Hyperlipidemia (plasma triglyceride concentration > 150mg/dl), Pregnancy, Hematocrit <34%

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-12-12 (Actual); Study Completion 2010-12-12 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 2-3 hours
  A hyperinsulinemic-euglycemic clamp will be used to assess insulin sensitivity.

SECONDARY OUTCOMES:
Resting Metabolic Rate | 20-30 min

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Michigan Clincal Research Unit, Ann Arbor, Michigan, United States